CLINICAL TRIAL: NCT01118975
Title: GCC 0845: Pilot and Phase II- Vorinostat and Lapatinib in Patients With Advanced Solid Tumor Malignancies and Women With Recurrent Local-Regional or Metastatic Breast Cancer to Evaluate Response and Biomarkers of EMT and Breast Cancer Stem Cells
Brief Title: GCC 0845:Vorinostat and Lapatinib in Advanced Solid Tumors and Advanced Breast Cancer to Evaluate Response and Biomarkers
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lost sponsorship for study drug
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: University of Maryland Greenebaum Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00040048
Record Dates: First submitted 2010-05-05; First posted 2010-05-07 (Estimated); Results first posted 2014-04-24 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-10

CONDITIONS: Breast Cancer; Neoplasm Metastasis
Keywords: lapatinib ditosylate; Zolinza (vorinostat); Cancer Stem Cells
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Vorinostat; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pilot Phase - Vornistat 200 to 400mg + Lapatinib (Experimental): lapatinib 1,250 mg continuous daily and escalating doses of vorinistat (200mg run-up, 300mg, and 400mg 4 days on 3 days off)
  Interventions: Drug: Vorinostat; Drug: Lapatinib
- Phase II - Vorinistat 400mg + Lapatinib (Experimental): lapatinib 1,250 mg continuous daily and vorinostat 400 mg 4 days on 3 days
  Interventions: Drug: Vorinostat; Drug: Lapatinib

INTERVENTIONS:
Drug: Vorinostat — 300 mg 4 days on then 3 days off
  As defined in the protocol, the dose of vorinostat was increased to 400 mg 4 days on then 3 days off in the pilot phase because the adverse event threshold was not met. In the Phase II cohort, the dose of vorinistat was 400 mg 4 days on and 3 days off.
  Other Names: Zolinza
Drug: Lapatinib — 1,250 mg once daily
  Other Names: Tykerb

SUMMARY:
This research is being done to find out how safe and how well the combination of lapatinib and vorinostat works against advanced cancers.

DETAILED DESCRIPTION:
Lapatinib is an anti-cancer drug that is approved by the Food and Drug Administration (FDA) for the treatment of metastatic HER2-positive breast cancer. HER2 is a protein involved in the growth of some cancer cells. In lab tests and small clinical studies, lapatinib is also found to kill other types of cancer that have another related protein called epidermal growth factor receptor (EGFR). For participants who have other cancers, the use of lapatinib in this study is investigational. This means the drug is not FDA approved for this use.

Vorinostat is only FDA approved for the treatment of cutaneous T cell lymphoma (a type of cancer). Vorinostat is not currently FDA approved for breast cancer or any other type of cancer. The use of vorinostat in this study is investigational.

Cancer cells can travel through the blood stream and spread to other organs. This process is called metastasis. Lab tests and small clinical trials have shown that vorinostat kills some cancer cells and prevents these cancer cells from traveling through the blood stream. These trials have shown that vorinostat improves how well lapatinib kills cancer cells.

Newer studies have also shown that a subset of cells, called "cancer stem cells," can come back, spread, and become resistant to the usual chemotherapy. In laboratory tests, we found that vorinostat and lapatinib can reduce the number of cancer stem cells. We are looking at combining vorinostat and lapatinib in the hope that we can reduce the number of cancer stem cells and cancer cells traveling through the blood stream.

There are two parts to this study.

First part- We want to learn more about the best dose of vorinostat to be given with lapatinib. We want to learn about how much vorinostat and lapatinib goes into the blood during treatment. We also want to learn the side effects (safety) of the combination of vorinostat and lapatinib. All patients will receive the FDA-approved dose of lapatinib. The first group of patients will get a slightly lower dose of vorinostat than is given normally. If the side effects are not too serious, the next group of patients will get the dose of vorinostat that is given normally.

Second part- We will find out how well the combination of vorinostat and lapatinib works in patients with HER2-positive metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2.
* Consent for peripheral blood sampling for analysis of circulating tumor cells.
* Patients must have adequate organ and marrow function as defined by the protocol.
* Female patients with histologically confirmed adenocarcinoma of the breast with recurrent local-regional disease, or metastatic disease that have progressed after treatment with regimens that include an anthracycline, a taxane, or trastuzumab.
* Human Epidermal growth factor Receptor 2 (HER2) positive in the primary or secondary tumor tissue as defined by:

  * Grade 3plus staining intensity (on a scale of 0 to 3) by means of Immunohistochemistry (IHC) analysis OR
  * Gene amplification on fluorescence in situ hybridization (FISH) greater than or equal to 2.2.
* Patients must have measurable disease by the Response Evaluation Criteria In Solid Tumors (RECIST)criteria at the time of enrollment.
* Prior trastuzumab therapy is allowed. Trastuzumab should be stopped at least 4 weeks prior to enrollment.

Exclusion Criteria:

* Patients receiving any other investigational agents.
* Prior exposure to lapatinib, vorinostat, or other Histone deacetylase (HDAC) inhibitors. Prior valproic acid exposure is allowed providing this is a greater than or equal to 30 days wash-out period.
* History of allergic reactions or hypersensitivity to compounds of similar chemical or biologic composition to vorinostat or lapatinib.
* Patients with history of clinically significant or uncontrolled cardiac disease, as defined by the protocol, or any significant cardiac condition that in the judgment of the investigator is unsuitable.
* Significant chronic or recent (less than 30 days) acute gastrointestinal disorder with diarrhea as a major symptom (e.g. Crohn's disease, malabsorption, or Grade 2 or greater diarrhea of any etiology at baseline).
* Prior exposure to more than 360 mg/m2 doxorubicin or liposomal doxorubicin, more than 120 mg/m2 mitoxantrone, or more than 90 mg/m2 idarubicin, or elevated baseline cardiac troponin T (more than upper limit of normal).
* Patients with active Central Nervous System (CNS) metastasis and/or carcinomatous meningitis are excluded. Patients with CNS metastasis who have completed a course of therapy would be eligible for the study provided they are clinically stable for 3 weeks prior to entry as defined as: (1) no evidence of new or enlarging CNS metastasis and (2) off steroids and/or anticonvulsants, for at least 4 weeks before an enrollment.
* Female patient that is pregnant or breastfeeding or expecting to conceive during the study. Women able to have children must have a negative pregnancy test prior to enrollment. All patients must use two effective methods of contraception (including a barrier method) during treatment and for 12 weeks after stopping treatment.
* The patient is known to be Human immunodeficiency virus (HIV), Hepatitis B, or Hepatitis C-positive (test results are not required in order to participate).
* Patients with current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirement.
* Previous or current systemic malignancy within the past 3 years other than the following: Female- breast cancer or adequately treated carcinoma in-situ of the cervix, or Female and Male- basal/squamous carcinoma of the skin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saranya Chumsri, MD, Principal Investigator — University of Maryland, College Park
Locations (1):
- University of Maryland Greenebaum Cancer Center, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pilot Phase - Vornistat 200 to 400mg + Lapatinib | Phase II - Vorinistat 400mg + Lapatinib
Started | 9 | 3
Completed | 9 | 2
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pilot Phase - Vornistat 200 to 400mg + Lapatinib | Phase II - Vorinistat 400mg + Lapatinib | Total
Number analyzed (Participants) | 9 | 3 | 12
Age, Customized [Median (Full Range); unit: years] | 52 [25 to 66] | 51 [42 to 66] | 52 [25 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 12
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicities
Description: Safety and tolerability were assessed. Adverse events and dose limiting toxicities were recorded during an escalting dose pilot phase.
Time Frame: 6 weeks
Measure: Number; unit: Dose limiting toxicities
Groups:
- Pilot Phase: The pilot phase consisted of an escalating dose design. Three patients received lapatinib 1,250 mg daily plus 300 mg vorinistat 4 days on then 3 days off. This dose was tolerated so six more patients recieved lapatinib 1,250 mg daily plus 400 mg vorinistat 4 days on 3 days off.
Arm/Group | Pilot Phase
Number analyzed (Participants) | 9
Dose limiting toxicities | 0

2. Primary Outcome: Clinical Benefit Rate
Description: The Clinical Benefit Rate is the number of patients with either Complete Response (CR), Partial Response (PR), or Stable Disease (SD) for ≥ 6 months
Time Frame: Radiological evaluations are performed every 12 weeks to determine disease status
Measure: Number; unit: participants
Groups:
- Phase II - Vorinistat 400mg + Lapatinib: lapatinib 1,250 mg continuous daily and vorinostat 400 mg 4 days on 3 days off
Arm/Group | Phase II - Vorinistat 400mg + Lapatinib
Number analyzed (Participants) | 3
participants | 1

ADVERSE EVENTS:
Arm/Group | Pilot Phase - Vornistat 200 to 400mg + Lapatinib | Phase II - Vorinistat 400mg + Lapatinib
Serious Adverse Events (participants affected / at risk) | 1/9 | 0/3
Other Adverse Events (participants affected / at risk) | 9/9 | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pilot Phase - Vornistat 200 to 400mg + Lapatinib (N=9) | Phase II - Vorinistat 400mg + Lapatinib (N=3)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Patient was hospitalized for upper respiratory infection. This event was deemed unrelated to the treatment
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Patient was hospitalized for dyspnea. This event was deemed to be unlikely to be related to study treatment.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pilot Phase - Vornistat 200 to 400mg + Lapatinib (N=9) | Phase II - Vorinistat 400mg + Lapatinib (N=3)
Fatigue (General disorders) | 3 (3) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (9) | 1 (3)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Anorexia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Skin Atrophy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Bony lesion (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dental abscess (Infections and infestations) | 1 (2) | 0 (0)
Depression (Psychiatric disorders) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 1 (3) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Ear ache (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Elevated chloride (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Elevated creatinine (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Elevated phosphorus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Elevated protein (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Elevated SGPT (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Elevated uric acid (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Headache (Gastrointestinal disorders) | 2 (3) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hot flashes (Endocrine disorders) | 2 (2) | 0 (0)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypertension (Cardiac disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 3 (5) | 0 (0)
Insomnia (General disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Migranes (General disorders) | 1 (1) | 0 (0)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Neuropathy (Nervous system disorders) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Ocular discharge (Eye disorders) | 1 (1) | 0 (0)
Pain - back, chest or shoulder (General disorders) | 3 (3) | 0 (0)
Pain - limbs (General disorders) | 3 (3) | 0 (0)
Prolonged QTc (Cardiac disorders) | 1 (1) | 0 (0)
Pruritis/itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Radiation dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (5) | 0 (0)
Skin nodules (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Thrush (Infections and infestations) | 1 (1) | 0 (0)
Weight loss (Metabolism and nutrition disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The most important limitation of this study is that the Phase II efficacy portion was terminated early by the sponsor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less